CLINICAL TRIAL: NCT01874106
Title: Effect of Anti-inflammatory Diet on Inflammatory, Oxidative and Nutritional Markers in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maryam Ekramzadeh, PhD (Other)
Collaborators: Shiraz University of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Maryam Ekramzadeh, PhD, PhD, Shiraz University of Medical Sciences
Organization: Shiraz University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 916425
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Inflammation; Malnutrition; Protein Energy Wasting Syndrome; Oxidative Stress; Diet Therapy
Keywords: Hemodialysis; Diet; Inflammation; Malnutrition
MeSH Terms: conditions — Inflammation; Malnutrition | interventions — Diet Therapy; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diet therapy (Experimental): The patients in this arm were educated to follow a especial type of diet (anti-inflammatory diet)in addition to nutrition counseling for 10 weeks.
  Interventions: Other: Diet Therapy
- Control Group (Other): The patients in this arm received nutrition counseling and education in general based on their needs as a control group for 10 weeks.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Diet Therapy — The patients in this arm were educated to follow a especial type of diet (anti-inflammatory diet)in addition to nutrition counseling for 10 weeks.
  Arms: Diet therapy
Other: Control Group — The patients in this arm received nutrition counseling and education in general based on their needs as a control group for 10 weeks.
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate the effect of especial diet therapy "Anti-inflammatory Diet" on inflammatory, oxidative stress, and nutritional markers in the context of protein-energy wasting syndrome(PEW) in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are on hemodialysis(HD) at least two times a week for 3months or more without any internment illness or admission

Exclusion Criteria:

* Hospitalization because of sepsis or surgery 3 months prior to intervention
* Cirrhosis
* Hepatitis virus infection
* Human Immunodeficiency virus infection
* Acquired Immunodeficiency Syndrome
* Active malignancy
* Active infection
* Absence of communication
* Mental Impairment
* Terminal illness
* Tube feedings
* Total parenteral nutrition
* Pregnancy
* Not previously seen by a dietitian within 3 months prior to enrollment in the study
* Not expected to be transplanted within 6 months after the enrollment in the study
* Absence of malnutrition from a cause other than end stage renal disease(ESRD)
* Psychiatric conditions, preventing adherence to intervention
* Consuming immunosuppressive drugs or taking antioxidant supplements including Vitamin E, Vitamin C, N-acetyl- cysteine (NAC), Pentoxifylline, Lipoic acid,Fish-oil extracts (omega-3 fatty acids), Soy extracts(isoflavones), Green-tea preparations, Pomegranate extracts, Grape extracts within 2 months prior to enrollment in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in serum Albumin | 10 weeks

SECONDARY OUTCOMES:
Change in Subjective Global Assessment (SGA) score | 10 weeks
Change in Malnutrition-inflammation score(MIS) | 10 weeks
Change in serum C-Reactive Protein(CRP) | 10 weeks
Change in serum malondialdehyde(MDA) | 10 weeks
Change in serum Interleukin-6(IL-6) | 10 weeks
Change in serum total antioxidant capacity(TAC) | 10 weeks
Change in serum ferritin | 10 weeks
Change in serum total iron binding capacity(TIBC) | 10 weeks
Change in serum urea nitrogen | 10 weeks
Change in serum creatinine | 10 weeks
Change in serum phosphorus | 10 weeks
Change in body fat mass index(BFMI) | 10 weeks
Change in fat free mass index(FFMI) | 10 weeks
Change in body cell mass(BCM) | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zohreh Mazloom, PhD, Study Director — Shiraz University of Medical Sciences, Faculty of Nutrition; Mohammadmahdi Sagheb, MD, Study Chair — Shiraz University of Medical Sciences, Nephrology Urology Research Center
Locations (1):
- Shiraz University of Medical Sciences, Department of Nutrition, Shiraz, Fars, Iran